CLINICAL TRIAL: NCT02703376
Title: Oral Prednisolone in the Treatment of Esophageal Stricture After Esophageal Surgery
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nagasaki University (Other)
Responsible Party: Principal Investigator, Kobayashi Shinichiro, Assistant professor, Nagasaki University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NagasakiU2
Record Dates: First submitted 2016-01-18; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Anastomotic Stricture
MeSH Terms: interventions — Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients after esophageal surgery (Other): Oral Prednisone for 12 weeks
  Interventions: Drug: Oral Prednisone

INTERVENTIONS:
Drug: Oral Prednisone — Intakes of Oral Prednisone for 12 weeks after balloon dilations
  Other Names: prednisolone

SUMMARY:
This study is safety and proof-of-concept study for oral prednisolone in the treatment of esophageal stricture after esophageal surgery. The patients who develop the severe esophageal strictures from 28 days after esophageal surgery are included. Primary outcomes are Safety and Success rate of this treatment.

DETAILED DESCRIPTION:
Esophageal strictures are common complications after surgery and aggressive endoscopic submucosal dissection (ESD) for early-stage esophageal cancer and adenocarcinoma. However, patients, who develop esophageal strictures after extensive operations, usually develop refractory strictures. Although there are several treatments for refractory strictures, their utility is limited.

Yamaguchi and colleagues have developed new treatments using oral prednisolone. They have shown the safety and potential efficacy to prevent esophageal strictures after ESD. However, the efficacy and safety of oral prednisolone is not evaluated to esophageal stricture after esophageal surgery.

This study is safety and proof-of-concept study for oral prednisolone in the treatment of esophageal stricture after esophageal surgery. The patients who develop the severe esophageal strictures from 28 days after esophageal surgery are included. Primary outcomes are Safety and Success rate of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients who develop the severe esophageal strictures from 28 days after esophageal surgery

Exclusion Criteria:

* Pulmonary and cardiac disorders
* Liver and renal dysfunctions
* Allergic
* Pregnancy
* infectious disease
* Unsuitable condition

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-03 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Clavien-Dindo Classification | for 12 weeks after the intervention
Incidence of Adverse Events of Grade 3 and Grade 4 of CTCAE v4.0 | for 12 weeks after the intervention
  physical conditions, clinical laboratory abnormalities, and ECG abnormalities
Incidence of treatment discontinuations, modifications, and interruptions due to adverse events | for 12 weeks after the intervention

SECONDARY OUTCOMES:
Rate of re-strictures at 85 postoperative days | for 12 weeks after the intervention
Number of participants with endoscopic classification of strictures before intervention | before the intervention
Dysphagia score | for 12 weeks after the intervention
Session of the dilatation | for 12 weeks after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kobayashi Shinichiro, Study Director — Department of Surgery Nagasaki University Graduate School of Biomedical Sciences
Locations (1):
- Nagasaki University, Nagasaki, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamaguchi N, Isomoto H, Nakayama T, Hayashi T, Nishiyama H, Ohnita K, Takeshima F, Shikuwa S, Kohno S, Nakao K. Usefulness of oral prednisolone in the treatment of esophageal stricture after endoscopic submucosal dissection for superficial esophageal squamous cell carcinoma. Gastrointest Endosc. 2011 Jun;73(6):1115-21. doi: 10.1016/j.gie.2011.02.005. Epub 2011 Apr 14. PMID 21492854
- [Background] Kobayashi S, Kanai N, Ohki T, Takagi R, Yamaguchi N, Isomoto H, Kasai Y, Hosoi T, Nakao K, Eguchi S, Yamamoto M, Yamato M, Okano T. Prevention of esophageal strictures after endoscopic submucosal dissection. World J Gastroenterol. 2014 Nov 7;20(41):15098-109. doi: 10.3748/wjg.v20.i41.15098. PMID 25386058